CLINICAL TRIAL: NCT06678880
Title: Chronobiological Basis of Depression During the Menopause Transition
Brief Title: Chronobiological Basis of Menopausal Depression: Correcting Misaligned Circadian Rhythms With Sleep and Light Interventions
Acronym: SALI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Barbara L. Parry, M.D., Professor of Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH134120
Record Dates: First submitted 2024-10-30; First posted 2024-11-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Depression; Depression During the Menopausal Transition; Menopausal Depression
Keywords: Menopause; depression; sleep and light intervention; melatonin; circadian rhythm; Chronobiology
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants assigned to the experimental condition.
  Interventions: Behavioral: Phase Advanced Intervention (PAI)
- Active Comparator Group (Active Comparator): Participants assigned to the active comparator condition.
  Interventions: Behavioral: Phase Delay Intervention (PDI)

INTERVENTIONS:
Behavioral: Phase Advanced Intervention (PAI) — Phase-advanced restricted sleep (i.e., sleep 9pm-1am only) for 1 night, followed by morning bright white light for 30 min/day for 2 weeks.
  Arms: Experimental Group
Behavioral: Phase Delay Intervention (PDI) — Phase-delayed restricted sleep (i.e., sleep 3am to 7am only) for 1 night, followed by evening bright white light for 30 min/day for 2 weeks.
  Arms: Active Comparator Group

SUMMARY:
The goal of this clinical trial is to learn more about mood, sleep, and activity during menopause. The main question it aims to answer is: can mood and sleep dysfunction in menopause be improved by resetting misaligned circadian rhythm through one night of strategic sleep timing adjustment and two weeks of exposure to bright light at a certain time of day? Researchers will compare sleep timing (earlier vs. later) and bright white light exposure (morning or evening) to investigate the effect of melatonin levels on mood, sleep, and activity. Participants will 1) submit urine samples to measure melatonin levels, 2) be assigned to advance or delay their sleep for one night, 3) sit in front of a light box for 30 minutes per day (morning or evening) for 14 days, 4) complete questionnaires about their mood and sleep, and 5) wear a device that will measure their activity.

DETAILED DESCRIPTION:
Significant hormonal changes during perimenopause (P-M) may disrupt circadian rhythm (CR), manifesting as mood, sleep and activity dysfunction, increasing depressive illness risk. In this proposal, the investigators aim to test further a hypothesis of CR dysregulation in P-M mood and sleep dysfunction by administering critically-timed sleep + light interventions (SLI) designed to target and correct CR misalignment, and thereby improve mood and sleep. By this approach, the investigators aim to optimize P-M health and prevent disease and disability.

Hypotheses are: 1) SLI which phase-advance (shift earlier) vs phase-delay (shift later) CRs, best measured by melatonin, will ameliorate mood and sleep dysfunction, and 2) A corrective phase-shift in the primary biological target, melatonin timing, will be a significant mediator of improved function. In P-M depressed participants (DP) vs normal controls (NC), the investigators recently reported increased plasma melatonin secretion and delayed morning melatonin offset associated with mood and sleep disturbances; correcting the phase-delayed melatonin CR with critically-timed sleep (wake therapy) + light interventions improved mood and sleep within 1-2 weeks, correlating significantly with melatonin phase-advance.

To confirm target engagement and intervention mechanisms, in P-M women the investigators will compare 1) an Active Phase-Advance Intervention (PAI): phase-advanced restricted sleep (sleep 9pm-1am) for 1 night, followed by 2 weeks of phase-advancing morning (AM) bright white light (BWL) for 30 min/day starting within 30 min of wake time, vs 2) a Control Phase-Delay Intervention (PDI): phase-delayed restricted sleep (sleep 3-7am) for 1 night, followed by 2 weeks of phase-delaying evening (PM) BWL for 30 min/day ending 30 min before bedtime. In pilot data, the investigators found relatively inert effects of Control PDI on melatonin and nonsignificant (non-worsening) effects on mood and sleep. Combining SLI hastens, potentiates and maintains their beneficial effects. In a randomized parallel design in 100 P-M women with mood and sleep/activity dysfunction, the investigators will administer either PAI or PDI at home (to enhance ecological validity), assessing effects on psychometric measures, urinary 6-sulfatoxy-melatonin (6-SMT) and actigraphy sleep/activity.

This innovative combination of SLI identifies novel targets for health and disease prevention and addresses an unmet therapeutic need in P-M women. It extends to the P-M our investigations of CR dysregulation and its restoration with SLI in other mood and sleep disorders associated with hormonal change in premenstrual and peripartum depression. This approach potentially offers a safe, efficacious, rapid-acting, well-tolerated, nonpharmacological, sustainable, affordable, home, and thus effective, intervention that can reduce health disparities. This work also forms the basis for future trials, aiming to optimize treatment outcomes by identifying chronobiological targets specific to an individual, the goal of personalized, preventative medicine.

ELIGIBILITY:
Inclusion Criteria:

* Perimenopausal women with irregular menstrual cycles for at least 3 months
* Above age 18
* Experiencing at least moderate depression symptoms (i.e., score of at least 10 on PHQ-9)

Exclusion Criteria:

* Actively suicidal or psychotic
* History of bipolar disorder
* Staring new medications that would affect outcome measures (e.g., melatonin)
* Those in whom sleep restriction would be ill-advised (e.g., patients with epilepsy or those with occupations whose safety would be compromised).
* Women whose body mass index (BMI) exceeds the NIH criteria of <18 or > than 30

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — As only biological women undergo menopause, only biological women will be eligible for this study.
Enrollment: 120 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Urine-based 6-sulfatoxymelatonin (6-SMT) | Baseline and after completing two-week intervention.
  Change in melatonin onset, offset, and acrophase.
Structured Interview Guide for the Hamilton Rating Depression Scale with Atypical Depression Supplement (SIGH-ADS) | Baseline and after completing two-week intervention; sustained at two weeks post intervention completion through three months post intervention completion.
  Clinicians rate change in mood on a numerical scale where 0= little/no symptoms and a higher number indicates increased symptoms or impairment.
Patient Health Questionnaire (PHQ-9) | Baseline and after completing two-week intervention; sustained at two weeks post intervention completion through three months post intervention completion.
  PHQ-9 assesses mood. Participants rate items on a scale of 0 to 3, where 0 = Not at all; 1 = Several days; 2 = More than half the days; 3 = Nearly every day.
Sleep Quality Rating (SQR) | Baseline and after completing two-week intervention; sustained at two weeks post intervention completion through three months post intervention completion.
  Participants will rate their sleep quality as well as whether they feel rested and alert using a slider scale. For this scale, lower value indicates better scores while higher values indicate worse scores.
Objective Measures of Sleep | Continuous monitoring from one week prior to baseline through one week post intervention completion.
  Change in sleep timing and duration (objectively measured via continuously worn MotionWatch device)
Objective Measures of Physical Activity | Continuous monitoring from one week prior to baseline through one week post intervention completion.
  Change in physical activity (objectively measured via continuously worn MotionWatch device)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Parry, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego Hillcrest Medical Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to directly share individual participant data (IPD) with other investigators. If such data is requested, the investigators will consider each request individually to determine whether sharing of IPD is appropriate or feasible. However, the investigators will be providing de-identified data to the National Institution for Mental Health Data Archive (NDA) throughout the duration of the study as required by NIH. This data will be available to other investigators after the conclusion of the study per the guidelines and restrictions established by the NDA.